CLINICAL TRIAL: NCT00851019
Title: Dance Dance Revolution (DDR) Exergaming in Adults With Type 2 Diabetes Mellitus
Brief Title: Dance Dance Revolution (DDR) in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles Drew University of Medicine and Science (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-08-2177
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Last update posted 2013-03-27 (Estimated); Status verified 2013-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Exercise; Video game; Type 2 diabetes; Dance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DDR (Experimental): "Dance Dance Revolution" (DDR) Exergaming
  Interventions: Behavioral: DDR
- Treadmill (Active Comparator): Treadmill exercise
  Interventions: Behavioral: Treadmill

INTERVENTIONS:
Behavioral: DDR — Ad libitum attendance to engage in "Dance Dance Revolution" (DDR) Exergaming, for a 3-month period
  Arms: DDR
Behavioral: Treadmill — Ad libitum attendance to engage in treadmill exercise, for a 3-month period
  Arms: Treadmill

SUMMARY:
Regular physical activity is important for the treatment of type 2 diabetes, but it is often not sustained for many reasons, including lack of interest. New video games that involve physical movement ("exergames") may help in this regard. This study will compare the "exergame" "Dance Dance Revolution" (DDR) with traditional treadmill exercise on blood sugar control among sedentary, overweight or obese adults with type 2 diabetes.

DETAILED DESCRIPTION:
This study is a randomized, controlled trial of a 3-month ad libitum program of the "exergame" "Dance Dance Revolution" (DDR) versus traditional treadmill exercise. Each group of subjects will be assessed at baseline, and then assigned exclusively to one of the two exercise modalities. Subjects will be free to attend exercise sessions in their assigned exercise modality at the exercise facility, at a frequency, duration and intensity of their own choosing with minimal staff supervision, for a period of exactly 90 days; adoption of new exercise programs outside of the study will be prohibited. Dosages of any concurrent medications will be maintained constant, and all subjects will receive standardized nutrition counseling.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 inclusive
* Diagnosed type 2 diabetes mellitus (by ADA diagnostic criteria) for at least 1 year
* On stable doses of oral anti-hyperglycemic medications for at least 3 months (i.e., sulfonylureas, metformin, thiazolidinediones, and/or DPP-4 inhibitors; GLP-1 analogues may also be permitted)
* Hemoglobin A1c level between 7.5% and 9.0% inclusive
* Body mass index (BMI) between 25.0 and 40.0 kg/m2 inclusive
* Able to engage in a regular program of mild-to-moderate intensity physical activity
* Subjects not currently engaged in any regimented exercise program outside of the usual activities of daily living that is intended to achieve metabolic changes (e.g., weight loss, athletic training, etc.)
* Able to give informed consent and cooperate with all necessary procedures of the study

Exclusion Criteria:

* Any contraindications to a regular program of mild-to-moderate intensity exercise, or any cardiovascular, pulmonary, orthopedic, rheumatological or neurological conditions that may, in the opinion of the investigators, interfere with the subject's optimal participation in a regular exercise program, interfere with the quality of the data collected from the subject, or make a regular exercise program potentially hazardous
* Diabetes mellitus currently being treated with insulin and/or pramlintide
* Screening fasting plasma glucose (FPG) 300 mg/dL or greater or symptoms of hyperglycemia (polyuria, polydipsia); screening FPG < 60 mg dL, or a history of symptomatic hypoglycemia averaging more than once per day; or any other history suggestive of erratic glucose control
* Screening fasting triglycerides 500 mg/dL or greater; or LDL-cholesterol 200 mg/dL or greater; screening blood pressure averaging 180 mm Hg or greater systolic or 100 mm Hg or greater diastolic
* Subjects currently engaged in any regimented exercise program outside of the usual activities of daily living that is intended to achieve metabolic changes (e.g., weight loss, athletic training, etc.); any such activities occurring on a sporadic basis may still disqualify the subject, depending upon its frequency, to be judged at the discretion of the PI. Subjects must maintain their usual occupational and other routine daily activities during the study at a reasonably constant level.
* Subjects who routinely engage in DDR, either at home or video game arcades; "occasional" participation in DDR may still disqualify the subject, depending upon the frequency of participation, to be judged at the discretion of the PI
* Changing doses of any concurrent medications that are known to alter the study's outcomes (e.g., oral anti-hyperglycemic agents, lipid-lowering agents, weight loss agents, anti-hypertensive agents, systemic glucocorticoids, thyroid medications, hormone replacement therapies, oral contraceptives, etc.) or the anticipated need to start any of these medications; such medications taken concurrently must remain at constant dosages throughout the study.
* Past history of clinically significant dysfunction of other organ systems (e.g., known hepatic disease or hepatic transaminase levels greater than 3X the upper limit of the normal range other than steatohepatitis; known renal dysfunction or creatinine level 1.5 mg/dL or greater; past history of malignancies excluding cutaneous basal cell carcinoma; known chronic infections including HIV, endocrinopathies such as untreated thyroid disease, adrenal disease, or pituitary dysfunction, etc.), or any recent surgeries that preclude regular exercise, in the opinion of the investigators
* Active hemolytic anemia, known hemoglobinopathies, or any other state of accelerated RBC turnover that may alter the accuracy of the HbA1c measurement
* Pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2009-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c change from baseline | 3 months

SECONDARY OUTCOMES:
Body mass index change from baseline | 3 months
Body composition change from baseline | 3 months
Fasting lipid profile change from baseline | 3 months
Blood pressure change from baseline | 3 months
Fasting plasma glucose change from baseline | 3 months
HOMA-IR index change from baseline | 3 months
Aerobic fitness change from baseline | 3 months
Mean daily caloric intake | 3 months
Mean total exercise time | 3 months
Mean exercise energy expenditure | 3 months
Behavioral questionnaires change from baseline | 3 months
All adverse events | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Hsia, MD, Principal Investigator — Charles Drew University of Medicine and Science
Locations (1):
- Charles Drew University of Medicine and Science, Los Angeles, California, United States